CLINICAL TRIAL: NCT00750412
Title: An Assessment of Voluntary Adolescent Mental Health Screening and Referral in a Children's Hospital Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCHMC 2008-0987
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Mental Health
Keywords: TeenScreen; Mental Health; Adolescent Mental Health; Social Work
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TeenScreen (Experimental)
  Interventions: Behavioral: TeenScreen Program
- Treatment As Usual (No Intervention)

INTERVENTIONS:
Behavioral: TeenScreen Program — Adolescents who are randomized into the TeenScreen program and their parent/guardian will receive post-screening information, a facilitated referral, and case management services from a research social worker.
  Arms: TeenScreen

SUMMARY:
The purpose of this study is to compare the TeenScreen intervention to usual care for adolescents who screen positive for mental health problems in a pediatric emergency department. It is anticipated that adolescents receiving the TeenScreen intervention will be more likely to attend a first session of outpatient mental health services within 60 days of the initial screening than those receiving the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 11 and 17 years old
* Medically stable and presenting with a non-psychiatric complaint
* English speaking
* Parent/guardian present for consent
* Insurance coverage by Medicaid
* Hamilton County residents
* Not currently receiving mental health treatment

Exclusion Criteria:

* Less than 11 years or greater than 17 years old
* Parent/guardian not present at time of visit
* Medically unstable
* Non-English speaking
* Insurance other than Medicaid
* Presenting complaint is a mental health problem
* Currently receiving mental health treatment

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Verified mental health service use through clinical administrative data | 60 days after the initial mental health screening

SECONDARY OUTCOMES:
Measurement of depressive symptoms and impairment of functioning utilizing the Center for Epidemiological Studies-Depressions Scale and Sheehan Disability Score | 60 days after the initial mental health screening

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Grupp-Phelan, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center Division of Emergency Medicine, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Grupp-Phelan J, McGuire L, Husky MM, Olfson M. A randomized controlled trial to engage in care of adolescent emergency department patients with mental health problems that increase suicide risk. Pediatr Emerg Care. 2012 Dec;28(12):1263-8. doi: 10.1097/PEC.0b013e3182767ac8. PMID 23187979
- See also: Columbia University TeenScreen Program — http://www.teenscreen.org